CLINICAL TRIAL: NCT02741037
Title: Unidas Por la Vida: A Healthy Lifestyle Intervention for High-risk Latina Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: AltaMed Health Services Corporation (Other); University of California, San Diego (Other)
Responsible Party: Principal Investigator, Dara Sorkin, Associate Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 20097225
Record Dates: First submitted 2016-03-31; First posted 2016-04-18 (Estimated); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Diabetes; Obesity; Overweight
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dyadic lifestyle intervention (Experimental): Mothers and daughters participate in the Unidas partner intervention together.
  Interventions: Behavioral: Dyadic lifestyle intervention; Other: Usual Care
- Individual lifestyle intervention (Experimental): Mothers participate in the Unidas intervention alone, without their related daughters. Unrelated daughters participate in the Unidas intervention alone without their related mothers.
  Interventions: Behavioral: Individual lifestyle intervention; Other: Usual Care
- Usual Care (Other): Mothers and daughters receive usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Dyadic lifestyle intervention — Dyadic lifestyle intervention: The dyadic behavioral lifestyle intervention was modeled after the Diabetes Prevention Program (DPP), and was adapted to make it more easily accessible to low-income Latinas. In addition, this intervention arm has a dyadic component to examine the effectiveness of mothers and daughters engaging in the lifestyle intervention together as partners. Participants also will receive usual care.
  Arms: Dyadic lifestyle intervention
Behavioral: Individual lifestyle intervention — Individual lifestyle intervention: The individual behavioral lifestyle intervention was modeled after the Diabetes Prevention Program, and was adapted to make it more easily accessible to low-income Latinas. Mothers participate in the Unidas intervention alone, without their related daughters. Unrelated daughters participate in the Unidas intervention alone without their related mothers. Participants also will receive usual care.
  Arms: Individual lifestyle intervention
Other: Usual Care — Usual Care: Mother and daughter participants will receive Usual Care.

SUMMARY:
Mexican American women have significantly elevated rates of obesity and type 2 diabetes. The proposed study tests a novel intervention that capitalizes on an existing important family dyad (mothers and their adult daughters) to foster clinically significant and long-lasting health behavior change. If found to effective, this intervention strategy has great potential to address health disparities in this, and other, at-risk populations.

DETAILED DESCRIPTION:
Approximately half of Mexican-American women report having a sedentary lifestyle, and nearly 78% are overweight or obese. Compared to women in all other ethnic groups, Mexican-American women have the highest lifetime risk of type 2 diabetes. The development of culturally appropriate lifestyle interventions for this population is an urgent priority, and the proposed study accordingly will investigate a novel dyadic intervention designed to improve health behaviors and promote weight loss in two at-risk members of the same family: mothers with type 2 diabetes and their overweight/obese adult daughters who are at risk for developing diabetes. The intervention, Unidas por la Vida (United for Life), capitalizes on the importance of the family in Latino culture to mobilize an existing family dyad as a source of mutual support that is likely to foster greater and longer-lasting health behavior change. The study builds on a successful pilot study (R34 DK083500) that established the feasibility and acceptability of this dyadic behavioral lifestyle intervention in a high-risk sample of Mexican-American family members who share a risk for diabetes and its complications. The 16-week intervention was modeled after the Diabetes Prevention Program (DPP), but was adapted for use with mother daughter pairs and to be community-based and, thus, more easily accessible to low-income Latinas. Preliminary data from the Unidas pilot study indicated that the dyadic intervention promoted significant weight loss. The proposed study extends the successful pilot study to: 1) target weight loss > 5% of baseline body weight and to foster maintenance using a tapered intervention, 2) add comparison groups that permit evaluation of the improvement uniquely associated with the partner intervention, and 3) assess theoretically derived mediators of the intervention. Participants (N=460 mother-adult daughter dyads) will be randomized into one of three conditions: 1) dyadic (mother-daughter) participation in a Unidas partner intervention (Arm 1); 2) individual participation (mothers alone; unrelated daughters alone) in a Unidas individual intervention (Arm 2); and 3) mother-daughter dyad in a usual care only condition (Arm 3).

ELIGIBILITY:
Inclusion Criteria:

Mothers:

1. Are Mexican-American
2. Are age 18 and older
3. Have a body mass index (BMI) between 25 kg/m2 and 43 kg/m2.
4. Are diagnosed with type 2 diabetes
5. Live within a 25 mile radius of your adult daughter
6. Are fluent in either Spanish or English as your primary language
7. Are able to understand and sign an informed consent

Adult daughters:

1. Are Mexican-American
2. Are age 18 and older
3. Have a body mass index (BMI) between 25 kg/m2 and 43 kg/m2.
4. Live within a 25 mile radius of your mother
5. Are fluent in either Spanish or English as your primary language
6. Are able to understand and sign an informed consent

Exclusion Criteria:

1. Are male
2. Have a visual or hearing impairment, documented psychiatric and/or life-threatening illness that precludes the ability to participate in a weight loss program and/or provide consent.
3. Are a mother with diabetes who is not able to start an exercise regimen or are likely to be injured (e.g., have uncontrolled high blood pressure).
4. Are pregnant or become pregnant during the course of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 710 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Longitudinal % change in body weight | 6, 12, and 18 months
  The study will compare longitudinal % change in body weight across the three study arms.

SECONDARY OUTCOMES:
Longitudinal change in dietary intake | 6, 12, and 18 months
  The study will examine whether changes in dietary intake are greatest among women in the partner intervention, compared to women in an individual intervention or in usual care, and to examine whether changes in dietary intake mediate the effects of the intervention on weight status and maintenance. Dietary intake will be measured with the Spanish version of the 2005 Block Food Frequency Questionnaire (FFQ). This instrument assesses portion sizes and frequency of consumption of over 100 food items, including foods selected for their cultural appropriateness for Mexican Americans to provide validated estimates of energy intake (total kilocalories) and macronutrient intake (including fat, carbohydrates and dietary fiber).
Longitudinal change in physical activity | 6, 12, and 18 months
  The study will examine whether changes in physical activity are greatest among women in the partner intervention, compared to women in an individual intervention or in usual care, and to examine whether changes in physical activity mediate the effects of the intervention on weight status and maintenance. The 7-day physical activity recall (PAR) will be used to assess physical activity at each study time point. Participants will be asked to estimate the number of hours spent each day (starting with the current day and working backwards) in sleep and in moderate, hard, and very hard physical activities.
Longitudinal change in interpersonal processes | 6, 12, and 18 months
  The study will examine whether changes in theoretically-derived mediating mechanisms, such as interpersonal processes, are greatest among women in the partner intervention, compared to women in the individual intervention or in usual care to examine whether changes in these processes mediate the effects of the intervention on dietary intake and in physical activity. Well-established methods of social network and social exchange assessment will be used to obtain detailed information about the involvement of participants' social network members in health-related social support, social control, and/or social undermining. Participants will be asked to identify social network members who have helped them make healthy lifestyle changes (social support), have prompted or urged them to do more to make such changes (social control), and/or have interfered (intentionally or unintentionally) with their efforts to make such changes (social undermining).
Longitudinal change in mother-daughter processes of mutual influence | 6, 12, and 18 months
  The study will examine actor-partner interdependence models to explore group differences in mother-daughter processes of mutual influence across the study arms, with this mutual influence expected to be greater and more strongly related to the primary and secondary outcomes for women in the partner intervention, compared to women in the individual intervention or in usual care.

CONTACTS AND LOCATIONS:
Overall Officials: Dara H Sorkin, Ph.D., Principal Investigator — University of California, Irvine; Karen S Rook, Ph.D., Principal Investigator — University of California, Irvine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorkin DH, Rook KS, Campos B, Marquez B, Solares J, Mukamel DB, Marcus B, Kilgore D, Dow E, Ngo-Metzger Q, Nguyen DV, Biegler K. Rationale and study protocol for Unidas por la Vida (United for Life): A dyadic weight-loss intervention for high-risk Latina mothers and their adult daughters. Contemp Clin Trials. 2018 Jun;69:10-20. doi: 10.1016/j.cct.2018.03.013. Epub 2018 Mar 26. PMID 29597006